CLINICAL TRIAL: NCT03809039
Title: A Randomised, Double-Blind, Placebo-Controlled Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of MT-6345 in Healthy Subjects
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of MT-6345 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Preclinical finding
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: MT-6345-E01; 2018-002478-39 (EudraCT Number)
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Results first posted 2021-09-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose: MT-6345 & Placebo (Experimental)
  Interventions: Drug: MT-6345; Drug: MT-6345 Placebo
- Multiple Ascending Dose: MT-6345 & Placebo (Experimental)
  Interventions: Drug: MT-6345; Drug: MT-6345 Placebo

INTERVENTIONS:
Drug: MT-6345 — MT-6345
Drug: MT-6345 Placebo — MT-6345 Placebo

SUMMARY:
The purpose of this study is to Investigate the Safety, Tolerability and Pharmacokinetics of MT-6345 in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

Additional screening criteria check may apply for qualification:

* Able to provide written informed consent to participate in this study after reading the participant information sheet and Informed Consent Form (ICF), and after having the opportunity to discuss the study with the Investigator or designee.
* Healthy and free from clinically significant illness or disease as determined by medical history, physical examination, laboratory and other tests at Screening and Day -1.
* A body weight of ≥60 kg for males and ≥50 kg for females and a body mass index (BMI) (Quetelet index) ranging from 18 to 30.0 kg/m2 inclusive at Screening and Day -1.
* In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the Protocol restrictions and requirements.

Exclusion Criteria:

Additional screening criteria check may apply for qualification:

* Subjects with clinically significant (in the opinion of the Investigator) endocrine, thyroid, hepatic, respiratory, gastrointestinal, neurological, renal, cardiovascular disease, or history (within the last 5 years) of any significant psychiatric/psychotic illness disorder (including anxiety, depression and reactive depression).
* Female subjects who are pregnant (positive pregnancy test at Screening or Day -1) or lactating.
* Having previously received MT-6345 as part of this study.
* Clinically relevant abnormal medical history, physical findings or laboratory values at Screening or Day -1 that could interfere with the objectives of the study or the safety of the subject, as judged by the Investigator.
* Subjects who test positive for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, human immunodeficiency virus (HIV)-1 or HIV-2 antibodies at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science,, Study Director — Tanabe Pharma America, Inc.
Locations (1):
- Investigational center, City Name, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects of Part 1 were selected for Part 2.
Groups:
- Part 1 and Part 2 Placebo; Part 1: MT-6345 1 mg; Part 1: MT-6345 5 mg; Part 1 and Part 2: MT-6345 20 mg; Part 1: MT-6345 60 mg; Part 1: MT-6345 120 mg; Part 1: MT-6345 240 mg: Single dose
- Part 3: Placebo; Part 3: MT-6345 60 mg: Multiple dose
Period: Part 1
Arm/Group | Part 1 and Part 2 Placebo | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1 and Part 2: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 3: Placebo | Part 3: MT-6345 60 mg
Started | 11 (11 subjects (2 subjects in each of Part 1 MT-6345 1 mg, 5 mg, 20 mg, 60 mg, 240 mg, and 1 subject in Part 1 MT-6345 120 mg) received a matching placebo per their respective dose. The subjects are unique subjects, and were not counted more than once across any arms except for Part 2 Placebo.) | 6 (The subjects are unique subjects, and were not counted more than once across any arms.) | 6 (The subjects are unique subjects, and were not counted more than once across any arms.) | 6 (The subjects are unique subjects, and were not counted more than once across any arms except for Part 2 MT-6345 20mg.) | 6 (The subjects are unique subjects, and were not counted more than once across any arms.) | 4 (The subjects are unique subjects, and were not counted more than once across any arms.) | 5 (The subjects are unique subjects, and were not counted more than once across any arms.) | 0 | 0
Completed | 10 | 6 | 6 | 5 | 6 | 4 | 5 | 0 | 0
Not Completed | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 and Part 2 Placebo | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1 and Part 2: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 3: Placebo | Part 3: MT-6345 60 mg
Started | 1 (2 subjects who received a matching placebo per Part 1 MT-6345 20mg were selected to return for Part 2. Out of 2 subjects, only 1 subject received the placebo, and another subject withdrew the consent after Part 1. Therefore, this 1 subject is not a unique subject and was not counted again in the total number of exposed subjects.) | 0 | 0 | 5 (6 subjects in Part 1 MT-6345 20mg were selected to return for Part 2. Out of 6 subjects, only 5 subjects received MT-6345, and 1 subject withdrew the consent after Part 1. Therefore, these 5 subjects are not a unique subject and were not counted again in the total number of exposed subjects.) | 0 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3
Arm/Group | Part 1 and Part 2 Placebo | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1 and Part 2: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 3: Placebo | Part 3: MT-6345 60 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (The subjects are unique subjects, and were not counted more than once across any arms.) | 6 (The subjects are unique subjects, and were not counted more than once across any arms.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6
Not completed — Withdrawn by study termination | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 6

BASELINE CHARACTERISTICS:
Population: The analysis population is the subjects of Part 1 and Part 3 since the subjects of part 2 were selected from part 1.
Groups:
- Part 1 Placebo; Part 1: MT-6345 1 mg; Part 1: MT-6345 5 mg; Part 1: MT-6345 20 mg; Part 1: MT-6345 60 mg; Part 1: MT-6345 120 mg; Part 1: MT-6345 240 mg: Single dose
- Part 3 Placebo; Part 3: MT-6345 60 mg: Multiple dose
- Total: Total of all reporting groups
Arm/Group | Part 1 Placebo | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 3 Placebo | Part 3: MT-6345 60 mg | Total
Number analyzed (Participants) | 11 | 6 | 6 | 6 | 6 | 4 | 5 | 2 | 6 | 52
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 11 | 6 | 6 | 6 | 6 | 4 | 5 | 2 | 6 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 11 | 6 | 6 | 6 | 6 | 4 | 5 | 2 | 6 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 6 | 6 | 6 | 6 | 4 | 5 | 2 | 6 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 11 | 6 | 6 | 6 | 6 | 4 | 5 | 2 | 6 | 52
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mild, Moderate and Severe Adverse Events
Description: The criteria of Mild, Moderate and Severe are as follows:
  Mild: The event is transient and easily tolerated by the subject.
  Moderate: The event causes discomfort and interferes with the subject's general condition.
  Severe: The event causes considerable interference with the subject's general condition and may be incapacitating.
Time Frame: Up to 6 weeks
Measure: Number; unit: participants
Groups:
- Part 2: Placebo; Part 2: MT-6345 20 mg: Single dose
Arm/Group | Part 1 Placebo | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: Placebo | Part 2: MT-6345 20 mg | Part 3: Placebo | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 11 | 6 | 6 | 6 | 6 | 4 | 5 | 1 | 5 | 2 | 6
participants
  Mild | 4 | 0 | 2 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 2
  Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MT-6345
Description: Cmax was measured for MT-6345 for the PK analysis set (PKPOP) subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: Part 1 and Part 2: Pre-dose and post-dose at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72 (Day 4), 120 (Day 6), 192 (Day 9), and 336 (Day 15 Follow-up Visit) hours. Part 3: Pre-dose and post-dose at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours.
Population: PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
ng/mL | 8.219 (1.414) | 37.37 (9.471) | 153.3 (38.85) | 386.2 (65.23) | 780.9 (118.5) | 1522 (301.7) | 141.0 (42.39) | 523.8 (200.7)

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of MT-6345
Description: Tmax was measured for MT-6345 for the PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Measure: Median (Full Range); unit: hour
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
hour | 0.75 [0.50 to 1.00] | 1.01 [1.00 to 1.52] | 1.00 [0.50 to 2.00] | 1.50 [0.50 to 2.01] | 1.50 [0.50 to 1.50] | 1.50 [1.00 to 1.50] | 2.00 [0.50 to 5.00] | 1.25 [0.50 to 2.00]

4. Secondary Outcome: Plasma Terminal Elimination Half Life (t½) of MT-6345
Description: t1/2 was measured for MT-6345 for the PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
hour | 34.89 (12.54) | 31.83 (7.16) | 34.99 (8.69) | 44.38 (10.76) | 46.03 (22.76) | 47.43 (31.58) | 39.46 (8.96) | 31.09 (8.69)

5. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to 24 Hours (AUC0-24h) of MT-6345
Description: AUC(0-24h) was computed for MT-6345 for the PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
ng.h/mL | 59.6 (12.6) | 342 (89.6) | 1350 (293) | 4050 (888) | 7570 (634) | 15100 (2830) | 1400 (288) | 4200 (938)

6. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Last Measurable Concentration (AUC0-last) of MT-6345
Description: AUC(0-last) was computed for MT-6345 for the PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
ng.h/mL | 115 (28.6) | 776 (284) | 3060 (1080) | 11100 (2590) | 21500 (8740) | 41200 (20100) | 3590 (1200) | 4200 (938)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-∞) of MT-6345
Description: AUC(0-∞) was calculated for the PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: Part 1 and Part 2: Pre-dose and post-dose at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 24, 48, 72 (Day 4), 120 (Day 6), 192 (Day 9), and 336 (Day 15 Follow-up Visit) hour. Part 3: Pre-dose and post-dose at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16 and 24 hours.
Population: PKPOP subjects in Part 1, Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
ng.h/mL | 126 (31) | 786 (285) | 3190 (1200) | 11200 (2640) | 21800 (9300) | 42200 (21200) | 3650 (1200) | 9570 (3530)

8. Secondary Outcome: Terminal Elimination Rate Constant (Kel) of MT-6345
Description: Kel was estimated for the PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: /h
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
/h | 0.0222 (0.0081) | 0.0226 (0.0044) | 0.0208 (0.005) | 0.0166 (0.005) | 0.0176 (0.0072) | 0.0198 (0.0104) | 0.0182 (0.0038) | 0.0244 (0.0096)

9. Secondary Outcome: Mean Residence Time (MRT) of MT-6345
Description: MRT was calculated for the PKPOP subjects in Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects in Part 1, Part 2 and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
hour | 42.1 (16.6) | 40.8 (10) | 43.9 (11.9) | 57.3 (14.5) | 58.3 (28.6) | 58.8 (40.6) | 50.3 (9.52) | 42.5 (11.9)

10. Secondary Outcome: Apparent Oral Clearance (CL/F) of MT-6345
Description: CL/F was measured for MT-6345 in the PKPOP subjects of Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects of Part 1, Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: litre per hour
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
litre per hour | 8.36 (1.93) | 6.89 (1.81) | 7.14 (2.93) | 5.79 (2.15) | 6.16 (2.15) | 7.30 (4.17) | 5.88 (1.60) | 6.92 (2.20)

11. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUC0-t) of MT-6345.
Time Frame: up to 2 weeks after dosing
Population: AUC0-t was not collected, and could not be assessed due to early study termination.
Arm/Group | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 0

12. Secondary Outcome: Apparent Volume of Distribution at Steady State (Vss/F) of MT-6345
Description: Vss/F was measured for MT-6345 in the PKPOP subjects of Part 1 and Part 2, and on Day 1 in Part 3.
Time Frame: as for outcome 2
Population: PKPOP subjects of Part 1, Part 2, and on Day 1 in Part 3.
Measure: Mean (Standard Deviation); unit: litre(s)
Arm/Group | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: MT-6345 20 mg | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 5 | 5 | 6
litre(s) | 335 (86.7) | 271 (60.3) | 286 (39.8) | 318 (82.4) | 314 (32.2) | 319 (85.5) | 284 (32.6) | 280 (82.4)

13. Secondary Outcome: Linearity Factor (LF) of MT-6345
Time Frame: up to 2 weeks after dosing
Population: LF was not collected, and could not be assessed due to early study termination.
Arm/Group | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 0

14. Secondary Outcome: Accumulation Ratio (RA) of MT-6345
Time Frame: up to 2 weeks after dosing
Population: RA was not collected, and could not be assessed due to early study termination.
Arm/Group | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 0

15. Secondary Outcome: Urinary Excreted Amount of Test Compound (Ae) of MT-6345
Description: Ae was measured for MT-6345 for the PKPOP subjects in Part 3.
Time Frame: Day 1 (0 hours to 24 hours) and Day 10 (0 hours to 24 hours)
Population: PKPOP subjects in Part 3.
Measure: Mean (Standard Deviation); unit: milligram(s)
Arm/Group | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6
milligram(s)
  Day 1 | 0.160 (0.0440)
  Day 10 | 0.255 (0.102)

16. Secondary Outcome: Urinary Excreted Amount of Test Compound Expressed as a Percentage of the Dose Administered (Ae%) of MT-6345
Description: Ae% was measured for MT-6345 for the PKPOP subjects in Part 3.
Time Frame: Day 1 (pre-dose and post-dose at 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12 and 16 hours) and Day 2 to Day 10 (pre-dose on each day)
Population: PKPOP subjects in Part 3.
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6
percentage of dose
  Day 1 | 0.3 (0.1)
  Day 10 | 0.4 (0.2)

17. Secondary Outcome: Renal Clearance (CLR) of MT-6345
Description: CLR was measured for MT-6345 for the PKPOP subjects in Part 3. For Day 10, CLR was not calculated because AUC(0-24h) on the last day of dosing was not calculated.
Time Frame: Day 1 (0 hours to 24 hours) and Day 10 (0 hours to 24 hours)
Population: PKPOP subjects in Part 3.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part 3: MT-6345 60 mg
Number analyzed (Participants) | 6
L/h | 0.0390 (0.0110)

ADVERSE EVENTS:
Time Frame: From the time written informed consent was obtained from a subject until the end of the Follow-up Period or the withdrawal from the study were recorded, up to 6 weeks.
Arm/Group | Part 1 Placebo | Part 1: MT-6345 1 mg | Part 1: MT-6345 5 mg | Part 1: MT-6345 20 mg | Part 1: MT-6345 60 mg | Part 1: MT-6345 120 mg | Part 1: MT-6345 240 mg | Part 2: Placebo | Part 2: MT-6345 20 mg | Part 3: Placebo | Part 3: MT-6345 60 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/5 | 0/1 | 0/5 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/6 | 0/6 | 0/6 | 0/6 | 0/4 | 0/5 | 0/1 | 0/5 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 4/11 | 0/6 | 2/6 | 1/6 | 2/6 | 1/4 | 2/5 | 0/1 | 2/5 | 0/2 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Placebo (N=11) | Part 1: MT-6345 1 mg (N=6) | Part 1: MT-6345 5 mg (N=6) | Part 1: MT-6345 20 mg (N=6) | Part 1: MT-6345 60 mg (N=6) | Part 1: MT-6345 120 mg (N=4) | Part 1: MT-6345 240 mg (N=5) | Part 2: Placebo (N=1) | Part 2: MT-6345 20 mg (N=5) | Part 3: Placebo (N=2) | Part 3: MT-6345 60 mg (N=6)
Medical device site reaction (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fungal skin infections (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03809039/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT03809039/SAP_001.pdf